CLINICAL TRIAL: NCT06823128
Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients with Severe Stenosis or Occlusion of Anterior Intracranial Circulation Vessels
Acronym: RICASO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RICASO
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Remote ischemic conditioning; anterior circulation; Acute Ischemic Stroke; Occlusion; stenosis
MeSH Terms: conditions — Ischemic Stroke; Bites and Stings; Constriction, Pathologic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIC group+Guideline-based therapy (Experimental): RIC is given twice a day with 200mmHg pressure.
  Interventions: Device: RIC; Other: Guideline-based therapy
- Sham group+Guideline-based therapy (Active Comparator): RIC is given twice a day with 60mmHg pressure.
  Interventions: Device: Sham; Other: Guideline-based therapy

INTERVENTIONS:
Device: RIC — Remote Ischemic Conditioning is given twice a day with 200mmHg pressure,last for 7 to 10 days.
  Arms: RIC group+Guideline-based therapy
Device: Sham — RIC is given twice a day with 60mmHg pressure, last for 7 to 10 days.
  Arms: Sham group+Guideline-based therapy
Other: Guideline-based therapy — Guideline-based therapy

SUMMARY:
The primary purpose of this study is to examine whether remote ischemic treatment can better the 90 - day neurological outcomes in acute ischemic stroke patients having severe stenosis or occlusion of anterior intracranial circulation vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18 years old or above.
2. Severe stenosis (70% - 99%) or occlusion of anterior intracranial circulation vessels, mainly including the intracranial segment of the internal carotid artery, middle cerebral artery (M1, M2) and anterior cerebral artery (A1, A2), which is confirmed by digital subtraction angiography (DSA), computed tomography angiography (CTA) or magnetic resonance angiography (MRA).
3. Patients with clinically diagnosed acute ischemic stroke who received remote ischemic treatment within 72 hours after the onset.
4. The NIHSS score ranges from 4 to 24.
5. The mRS score before stroke is less than or equal to 1.
6. informed consent.

Exclusion Criteria:

1. Patients with vessel recanalization after mechanical thrombectomy (TICI grade ≥ 2b).
2. Patients planning to receive intracranial endovascular treatment within 3 months.
3. Patients with cardiogenic embolism considered as the cause, such as rheumatic mitral or aortic valve stenosis, artificial heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, left ventricular wall thrombus or valvular vegetations, congestive heart failure, bacterial endocarditis, etc.
4. Patients diagnosed with acute posterior circulation cerebral infarction.
5. Symptoms caused by non - culprit vessels.
6. Ipsilateral extracranial vessel stenosis ≥ 70%.
7. Systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg, and uncontrollable by antihypertensive drugs.
8. Intracranial tumors, arteriovenous malformations or aneurysms.
9. Cerebral venous thrombosis or stenosis.
10. Any intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural) within 90 days before enrollment.
11. Severe coagulation abnormalities.
12. Any contraindications to remote ischemic conditioning: severe soft tissue injury, fracture or vascular injury of the upper limb, perivascular lesions of the distal upper limb, etc.
13. Patients with any serious diseases and a life expectancy of less than 1 year.
14. Patients who participated in other clinical trials within 3 months before enrollment or are currently participating in other clinical trials.
15. Patients who cannot be followed up (such as those without a fixed residence, overseas patients, etc.).
16. Pregnant or lactating women.
17. Patients who have previously received remote ischemic treatment or similar treatments.
18. Patients whom the researchers consider unsuitable for this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Distribution of 90-day mRS scores | 90±14 days after procedure
  The Modified Rankin Scale (mRS) measures degree of disability/dependence after a stroke, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death

SECONDARY OUTCOMES:
Distribution of 360-day mRS scores (to be analyzed separately in the subsequent study) | 90±14 days after procedure
  The Modified Rankin Scale (mRS) measures degree of disability/dependence after a stroke, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death
Proportion of patients with functional independence outcome (mRS 0-1) at 90-day | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Proportion of patients with functional independence outcome (mRS 0-2) at 90-day | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Proportion of patients with functional independence outcome (mRS 0-3) at 90-day | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
The proportion of early neurological deterioration | 7 (± 1 day) after procedure
  It is defined as an increase of ≥ 2 points in the NIHSS score on the 7th day compared to the baseline (excluding intracerebral hemorrhage).
Activities of Daily Living of Participants Assessed by Bathel Index at 90-day | 90 (± 14 days) after procedure
  10 rating items, each of which is categorized into 2-3 out of 5 levels: Unable, Needs major help, Needs help, Needs minor help, and Independent, and each item has a different score for each level. Independence was positively correlated with the final score.
Activities of Daily Living of Participants Assessed by Bathel Index at 360-day | 360(± 14 days) after procedure
  10 rating items, each of which is categorized into 2-3 out of 5 levels: Unable, Needs major help, Needs help, Needs minor help, and Independent, and each item has a different score for each level. Independence was positively correlated with the final score.
Incidences of adverse cardiovascular and cerebrovascular events, and recurrent ischemic events | 360 (± 14 days) after procedure
  Adverse cardiovascular and cerebrovascular events include myocardial infarction, heart failure, severe arrhythmia, cerebral infarction, cerebral hemorrhage, transient ischemic attack (TIA), and recurrent ischemic events include recurrent myocardial infarction and recurrent cerebral infarction.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, China

IPD SHARING:
Plan to Share IPD: No